CLINICAL TRIAL: NCT00727428
Title: Immunogenicity and Safety Study of GSK Biologicals' Trivalent Split Virion Influenza Vaccine Fluviral®, Thimerosal-free (FluLaval® TF), in Adults 18 to 60 Years of Age.
Brief Title: Immunogenicity and Safety of GSK Biologicals' FluLaval® TF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112219
Record Dates: First submitted 2008-08-01; First posted 2008-08-04 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: FluLaval® TF; Safety; Immunogenicity; Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: FluLaval® TF

INTERVENTIONS:
Biological: FluLaval® TF — One IM injection.

SUMMARY:
The present study is intended to assess a novel formulation of FluLaval. The idea is to obtain preliminary data on the safety and immune response to the FluLaval TF influenza vaccine in adults. These data will serve as a basis for further studies involving different populations. This protocol posting deals with objectives & outcome measures of the primary phase/study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol
* Male and female adults, 18 to 60 years of age.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination (stable health status with no exclusionary medical or psychiatric conditions).
* Access to a consistent means of telephone contact, which may be either in the home or at workplace, land line or mobile, but not a pay phone or other multiple-user device.

Exclusion Criteria:

* Acute disease at the time of enrollment.
* Significant acute or chronic, uncontrolled medical or psychiatric illness. "Uncontrolled" is defined as:

  * Requiring institution of new medical or surgical treatment within 1 month prior to study enrollment, or
  * Requiring the re-institution of a previously discontinued medication or medical treatment within one month prior to study enrollment, or
  * Requiring a change in medication dosage in the one month prior to study enrollment due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or
  * Hospitalization or an event fulfilling the definition of a SAE within 1 month prior to study enrollment.
* Any confirmed or suspected immunosuppressive condition including:

  * History of human immunodeficiency virus (HIV) infection,
  * Cancer or treatment for cancer, within 3 years of study enrollment.
* History of renal impairment.
* History of hepatic dysfunction due to hepatitis B, C or toxins including alcohol.
* Complicated insulin-dependent diabetes mellitus.
* Unstable cardiopulmonary disease requiring chronic medical therapy or associated with functional impairment.
* Presence of blood dyscrasias, including hemoglobinopathies and myelo- or lymphoproliferative disorder.
* Receipt of systemic glucocorticoidswithin 1 month of study enrollment, or chronic use of any cytotoxic or immunosuppressive drugs within six months of study enrollment. Inhaled and topical steroids are allowed.
* History of any demyelinating disease including Multiple Sclerosis and Guillain-Barré syndrome.
* Presence of an active neurological disorder.
* History of chronic alcohol consumption and/or drug abuse.
* Any significant disorder of coagulation that increases the risk of intramuscular injections or treatment with coumadin derivatives or heparin
* Receipt of an influenza vaccine during the 2007-8 influenza immunization season.
* Administration of any vaccines within 30 days prior to study enrollment or during the study period. Subjects who receive such treatment after enrollment will be followed per protocol and included in the safety analysis, but excluded from the according-to-protocol cohort.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the vaccination or planned use during the study period.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or planned during the study.
* Any known or suspected allergy to any constituent of FluLaval and/or any flu vaccines and/or history of anaphylactic-type reaction to consumption of eggs.
* A history of severe adverse reaction to a previous influenza vaccination.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for the duration of the study.
* Lactating/nursing female.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2008-08-05 (Actual); Primary Completion 2008-08-29 (Actual); Study Completion 2009-02-17 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) of hemagglutination inhibition (HI) antibody against each of the 3 vaccine influenza strains | Days 0 and 21
Seroconversion Rates (SCR) | Day 21
Seroprotection Rates (SPR) | Days 0 and 21
Seroconversion Factors (SCF) | Day 21

SECONDARY OUTCOMES:
Occurrence, intensity and investigator's assessment of relationship to vaccine of solicited local and general signs and symptoms | During the 4-day follow-up period after vaccination.
Occurrence, intensity, and investigator's assessment of relationship to vaccine of unsolicited local and general signs and symptoms | During the 21-day follow-up period after vaccination.
Occurrence, intensity and investigator's assessment of relationship to vaccine of SAEs and medically attended events | During the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

REFERENCES:
- See also: Results for study 112219 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/112219?search=study&#rs